CLINICAL TRIAL: NCT05431335
Title: Investigation of the Efficacy of Structured Exercise Program in Tension-Type Headache
Brief Title: Exercise Treatment in Tension Type Headache
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Munzur University (Other)
Responsible Party: Principal Investigator, Kubra Sagır, Research Assistant, PhD student, Munzur University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KubraTTH2022
Record Dates: First submitted 2022-06-14; First posted 2022-06-24 (Actual); Last update posted 2023-08-23 (Actual); Status verified 2023-08

CONDITIONS: Tension-Type Headache
Keywords: Exercise; Aerobic exercise; Structured exercise; Tension-type headache; Quality of life
MeSH Terms: conditions — Tension-Type Headache; Motor Activity

STUDY DESIGN:
Intervention Model Description: Parallel design randomized clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Structured exercise program (Experimental): The structured exercise program will be applied for 12 weeks, 2 days a week, for 45 minutes by a physiotherapist.
  Interventions: Other: Structured exercise program
- Aerobic exercise program (Other): The aerobic exercise program will be applied for 12 weeks, 2 days a week, for 45 minutes by a physiotherapist.
  Interventions: Other: Aerobic exercise program

INTERVENTIONS:
Other: Structured exercise program — It consists of aerobic exercise combined with breathing, strengthening exercises, and stretching exercises. Aerobic exercise will be performed similarly to the other group, only consisting of a five-minute warm-up period and a 15-minute aerobic load period.
  Strengthening exercises consist of deep cervical flexor muscles and shoulder region resistive exercises. Each exercise will be repeated as 15 repetitions, 2 sets.
  Stretching exercises are neck region stretching exercises. Each exercise will be performed with 10 seconds of stretching and 5 repetitions.
  Arms: Structured exercise program
Other: Aerobic exercise program — Aerobic exercise intensity will be determined by the Perceived Fatigue Scale (Borg scale). It consists of a ten-minute warm-up period (Borg 11), a 15-minute aerobic load (Borg 13-14), and a five-minute cool-down period(Borg 11). The warm-up and cool-down periods include brisk walking combined with breathing, and calisthenic exercises involving the upper and lower extremities; the loading period consists of exercises using a step-dance board accompanied by music. The number of repetitions will be increased progressively to keep the exercise intensity constant.
  Arms: Aerobic exercise program

SUMMARY:
Tension-type headache (TTH) is a common type of headache. Its incidence in women has been reported as 18%. It is thought to be associated with stress, contractions in peripheral muscles, and changes in pain transmission and inhibition mechanisms in the central nervous system. As a chronic pain, it can cause a decrease in the quality of life and work capacity, and significant disabilities in daily living activities and functions of the person.

Exercise treatments are one of the non-pharmacological methods in the management of TTH. Exercise reduces pain by activating descending inhibitory pathways, reducing stress response, increasing relaxation and oxygenation, and thus provides healing. By this mechanism, the effects of aerobic exercise programs on pain severity, depression, and quality of life in migraine and TTH have been demonstrated. One of the underlying causes of TTH is head-forward posture, causing ischemia, increased muscle tone, and abnormal loads in the upper cervical region. Therefore, cervical region strengthening and deep cervical flexor stabilization exercises also have an effect on TTH. Although it has been shown in the literature that different types of isolated exercise are superior to control groups in TTH, there is a need for higher quality studies showing the effect of exercise. There is a lack of evidence on the feasibility and effectiveness of combined exercise programs. It is thought that additional benefits can be obtained by using exercise types in combination in order to focus on the central and peripheral mechanisms of TTH. The effects of a structured exercise program in which aerobic, strengthening, and stretching exercises are used together are intriguing. The aim of our study is to determine the effects of the structured exercise program and whether it is superior to isolated aerobic exercises. Our study will also provide evidence to the literature on the effects of aerobic exercise programs.

64 volunteer patients who were diagnosed with chronic TTH in the neurology outpatient clinic and met the inclusion criteria will be included. Participants will be included in one of the structured exercise programs and aerobic exercise programs. Both exercise programs are planned for 12 weeks, 2 days a week for 45 minutes. Participants will be evaluated with outcome scales before and after exercise programs.

ELIGIBILITY:
Inclusion Criteria:

* Having a diagnosis of chronic TTH according to the criteria of the International Headache Society (ICHD-III beta version, 2013)
* If using antidepressant medication, to start using medication 2 months before participating in the study.
* not having a communication difficulty or problem,

Exclusion Criteria:

* Having heart disease, cardiac arrhythmia, cardiovascular disease
* Receiving chemotherapy, radiotherapy with malignancy and causing malignancy
* Having any neurological or orthopedic disorder that will disrupt the balance
* being pregnant
* Being addicted to alcohol and drugs
* Having a history of Disc herniation, Radiculopathy, and Surgery in the cervical region
* Increase in pain severity during treatment sessions
* Not attending more than three treatment sessions

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 64 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-10 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Change in pain-related quality of life | 1- a day before the exercise program 2-at the midst of treatment (and of the 8 weeks exercise) 3-at the time of discharge (end of the 12 weeks exercise program)
  It will be measured by the headache impact test (HIT-6). It provides quantitative information about migraine and headache, based on the patient's self-report. The scale consists of six items and questions pain severity, loss of work and leisure activity, fatigue, and cognitive characteristics. The score range of the scale is 36-78. As a result, ≤49 points are considered as no effect, 50-55 as moderately affected, 56-59 as markedly affected, and ≥60 as severely affected. Its validity and reliability study was maden.

SECONDARY OUTCOMES:
Change in pain severity | 1- a day before the exercise program 2- and of the 4 weeks of exercise, 3- and of the 8 weeks of exercise, 4-at the time of discharge (end of the 12 weeks exercise program)
  The pain severity will be evaluated using a 0-10 point visual analog scale (VAS). It will be evaluated with a pain diary every weeks.
Change in pain frequency | 1- a day before the exercise program 2- and of the 4 weeks of exercise, 3- and of the 8 weeks of exercise, 4-at the time of discharge (end of the 12 weeks exercise program)
  Pain frequency will be followed up with a pain diary during the 8-week treatment period.
Change in Pain duration, | 1- a day before the exercise program 2- and of the 4 weeks of exercise, 3- and of the 8 weeks of exercise, 4-at the time of discharge (end of the 12 weeks exercise program)
  Pain duration will be followed up with a pain diary during the 8-week treatment period.
Change in Amount of painkiller use | 1- a day before the exercise program 2- and of the 4 weeks of exercise, 3- and of the 8 weeks of exercise, 4-at the time of discharge (end of the 12 weeks exercise program)
  Use of painkillers will be followed up with a pain diary during the 8-week treatment period.
Change in Pressure pain threshold | 1- a day before the exercise program 2-at the midst of treatment (and of the 8 weeks exercise) 3-at the time of discharge (end of the 12 weeks exercise program)
  Trapezius, levator scapula, suboccipital, pectorals, and deltoid muscles will be evaluated with palpation, trigger point pressure pain threshold will be measured with an dolorimeter.
Change in Pain-related disability | 1- a day before the exercise program 2-at the midst of treatment (and of the 8 weeks exercise) 3-at the time of discharge (end of the 12 weeks exercise program)
  It will be evaluated with the Pain Disability Index. The scale is a simple and fast tool used to measure the limitation of daily functions due to pain in patients with chronic pain. It consists of a total of 7 parameters: family and home responsibilities, entertainment, social activity, profession, sexual life, self-care and daily life activities. The lowest score that can be obtained from the scale is 0, and the highest score is 70. A high score indicates a high disability level.
Change in cervical flexor muscle activation score | 1- a day before the exercise program 2-at the midst of treatment (and of the 8 weeks exercise) 3-at the time of discharge (end of the 12 weeks exercise program)
  Cranio-cervical Flexion Test will be used to evaluate cervical flexor muscle strength. It will be evaluated with the Cranio-cervical Flexion Test. The test evaluates the activation and isometric endurance of the deep cervical flexor muscles. The test will be evaluated with the stabilizer pressure biofeedback device developed by Physiotherapist Gwendolen Jull. It is the minimal pressure score measured.
Change in cervical flexor muscle performance index | 1- a day before the exercise program 2-at the midst of treatment (and of the 8 weeks exercise) 3-at the time of discharge (end of the 12 weeks exercise program)
  Cranio-cervical Flexion Test will be used to evaluate cervical flexor muscle strength. It will be evaluated with the Cranio-cervical Flexion Test. The test evaluates the activation and isometric endurance of the deep cervical flexor muscles. The test will be evaluated with the stabilizer pressure biofeedback device developed by Physiotherapist Gwendolen Jull. It is obtained by calculating all the contractions the participant was able to achieve.
Change in Proprioception | 1- a day before the exercise program 2-at the midst of treatment (and of the 8 weeks exercise) 3-at the time of discharge (end of the 12 weeks exercise program)
  The sense of cervical proprioception will be measured. "Head repositioning" targeting the neutral position of the head and "target angle tests" targeting 20˚ extension, 30˚ flexion, 30˚ lateral flexion and 30˚ rotation angles of the neck will be measured.
Change in Craniovertebral angle | 1- a day before the exercise program 2-at the midst of treatment (and of the 8 weeks exercise) 3-at the time of discharge (end of the 12 weeks exercise program)
  It will be used to measure cervical posture. For the craniovertebral angle measurement, the angle between the horizontal plane and the line drawn over the tragus and cervical 7th spine is measured.
Change in cervical region posture | 1- a day before the exercise program 2-at the midst of treatment (and of the 8 weeks exercise) 3-at the time of discharge (end of the 12 weeks exercise program)
  PostureScreen Mobile® app (PostureCo; http://postureanalysis.com/mobile/) will be used to measure head, neck and shoulder posture.The application has been shown to be valid and reliable for posture assessment. With the application, the angular values of the patient's posture are automatically created by taking the image of the patient from the front and both lateral sides.
Change in Exercise capacity | 1- a day before the exercise program 2-at the midst of treatment (and of the 8 weeks exercise) 3-at the time of discharge (end of the 12 weeks exercise program)
  It will be evaluated with the Six Minute Walk Test, which is a submaximal exercise test. After walking for 6 minutes on a 20 or 30 meter track in a straight corridor, the total distance walked is recorded in meters.
Change in Anxiety and depression | 1- a day before the exercise program 2-at the midst of treatment (and of the 8 weeks exercise) 3-at the time of discharge (end of the 12 weeks exercise program)
  It will be evaluated with The Hospital Anxiety and Depression Scale. The scale consists of 7 anxiety and 7 depression questions answered with a four-point Likert scale. As a result of the validity and reliability study, cut-off scores were found to be 10/11 for the anxiety subscale and 7/8 for the depression subscale.

CONTACTS AND LOCATIONS:
Overall Officials: Kübra Sağır, PhD student, Principal Investigator — Munzur University
Locations (1):
- Munzur Üniversity, Tunceli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Effect of manual therapy techniques on headache disability in patients with tension-type headache. Randomized controlled trial. — http://europepmc.org/article/med/24785463